CLINICAL TRIAL: NCT06854796
Title: Prospective, Multicentre, Randomized, Blind, Parallel-controlled Clinical Trial Evaluating the Efficacy and Safety of Recombinant Collagen Gel for Correcting Moderate to Severe Nasolabial Wrinkles
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shaanxi Giant Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XG2412
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Nasolabial Fold Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recombinant collagen coagulation glue (Experimental): The recombinant collagen gel produced by Shaanxi Juzi Biotechnology Co., Ltd. was used for 1-2 injections.
  Interventions: Device: Recombinant collagen gel
- collagen implant agent (Active Comparator): Treated with 1-2 injections of collagen implants for the treatment of nasolabial folds manufactured by Shuangmei Biotechnology Co., Ltd.
  Interventions: Device: collagen implant agent

INTERVENTIONS:
Device: Recombinant collagen gel — The test device uses a recombinant collagen gel developed by Shaanxi Juzi Biotechnology Co., Ltd., which is different from other designs. The main components of recombinant collagen gel are recombinant collagen, disodium hydrogen phosphate, potassium dihydrogen phosphate, sodium chloride, water for injection, after the injection, collagen can occupy a place at the injection site to improve the visual aging caused by soft tissue loss, wrinkles and depressions, and the special manufacturing process can ensure that the gel has smoothness and ductility, which helps to achieve a smooth and natural appearance, effectively and gradually improve wrinkles and plump cheeks.
  Arms: Recombinant collagen coagulation glue
Device: collagen implant agent — 1. After the product is injected into the skin, the collagen implant forms a soft mesh structure through condensation, which can make up for skin defects. 2. After implantation of this product, the connective tissue cells around the implantation site will grow into the collagen network structure and gradually form a bionic structure similar to normal tissue. 3. This product is absorbable and degradable. The collagen implant will be gradually decomposed by protease in the body, and the pressure, elongation and hierarchy of the implant site tissue will affect the final degradation and duration.
  Arms: collagen implant agent

SUMMARY:
Trial name: Prospective, multicentre, randomized, blind, parallel-controlled clinical trial to evaluate the efficacy and safety of recombinant collagen gel for correcting moderate to severe nasolabial wrinkles Sponsor: Shaanxi Juzi Biotechnology Co., LTD Objective: To evaluate the efficacy and safety of recombinant collagen gel prepared by Shaanxi Juzi Biotechnology Co., LTD Experimental design: A prospective, multicenter, randomized, blind, parallel controlled experimental design was adopted, and the comparison type was non-inferiority test Sample size: 244 cases Experimental group: control group =1:1 Scope of application: It is suitable for injection into facial dermis or subcutaneous tissue to correct moderate and severe nasolabial wrinkles Case selection: Inclusion criteria (1) Age 18-65 years old (including the threshold value), male and female; (2) Those who have a need to improve nasolabial wrinkles and are rated moderate or severe (corresponding to a score of 3 or 4) on the bilateral nasolabial Wrinkles Severity Rating Scale (as assessed by blind investigators); (3) Voluntarily participate in this clinical trial and sign the subject informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-65 years old (including threshold), regardless of gender;
2. There is a need to improve nasolabial folds, and the bilateral nasolabial folds severity rating scale (WSRS) is rated as moderate or severe (corresponding to a score of 3 or 4) by blinded researchers;
3. Voluntarily participate in this clinical trial and sign the informed consent form for the subjects.

Exclusion Criteria:

1. Patients with acute or advanced skin diseases (vitiligo, psoriasis, eczema, etc.), obvious scars, active inflammation, infections (bacterial, fungal, viral), cancerous or precancerous lesions, or unhealed wounds in the nasolabial groove area;
2. Those who have received permanent or semi permanent dermal filler treatment (such as hydroxyapatite calcium, polymethyl methacrylate, organosilicon, expanded polytetrafluoroethylene, etc.) at the folds of the nasolabial groove, or plan to receive filler treatment during the study period;
3. Screening for individuals who have undergone facial plastic surgery or other cosmetic procedures at the intended injection site or lower middle part of the nasolabial fold in the previous 6 months, which may affect the WSRS rating (such as facial lifting surgery, botulinum toxin injection, etc.); Or those who plan to undergo any other facial surgery, medication, or laser treatment during the study period;
4. Individuals who have received temporary filler injections such as cross-linked hyaluronic acid, collagen, or polylactic acid in the nasolabial groove area within the previous 12 months, or who have received non cross-linked sodium hyaluronate injections in the nasolabial groove area within the previous 6 months;
5. Scar lumps, scar constitution, and individuals in the active phase of infectious diseases;
6. Those who have bleeding tendency and used anticoagulants within 2 weeks (heparin, warfarin, sodium citrate, aspirin, etc.), uncontrolled diabetes (HbA1c ≥ 7.5%), malignant tumors and other serious systemic diseases, or autoimmune diseases, such as rheumatism, lupus erythematosus, or immune dysfunction;
7. Patients with platelet count below 50 × 109/L or abnormal coagulation mechanism (such as APTT ≥ 1.5 times the upper limit of normal) during the screening period;
8. Abnormal liver and kidney function during the screening period (AST, ALT>1.5 times the upper limit of normal values or Cr>1.5 times the upper limit of normal values);
9. Individuals who have a history of allergies or allergies to local anesthetics such as pig derived materials or collagen materials, potassium dihydrogen phosphate, disodium hydrogen phosphate, or lidocaine (allergic to one or more substances);
10. Visual impairment that affects the subject's self-evaluation;
11. Individuals with a history of psychological disorders and mental illnesses who are unable to cooperate during the trial period;
12. Pregnant or lactating women, and those planning to conceive during the trial period;
13. Individuals who have participated in clinical trials of other intervention devices or within 5 half lives of their last medication in a drug clinical trial within one month prior to the start of this trial;
14. Researchers believe that participants should not participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Effective rate of correcting and improving nasolabial folds 90 days after the last injection | 90 days ± 7 days after the last injection
  Evaluation method: Blind researchers trained in the Wrinkle Severity Rating Scale (WSRS) were used to grade the injection site photos of subjects before and after injection.
  Evaluation criteria: Compared with the screening period, if the severity score of bilateral nasolabial folds is reduced by at least one level 90 days after the last injection, it is considered effective improvement. Otherwise, it is considered ineffective improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- The Seventh Medical Center of the Chinese People's Liberation Army General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No